CLINICAL TRIAL: NCT02479438
Title: Gastroesophageal Reflux Disease Prospective Registry
Acronym: GERD
Status: Terminated | Type: Observational
Why Stopped: The study was terminated by the Principal Investigator's to redesign it using more efficient processes.
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 014-008
Record Dates: First submitted 2015-05-07; First posted 2015-06-24 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (1):
- Diagnosed with GERD: Collect data on GERD patients
  Interventions: Other: Diagnosed with GERD

INTERVENTIONS:
Other: Diagnosed with GERD — Recording of patient outcomes

SUMMARY:
The purpose of this registry is to evaluate information to determine which operations and treatments for gastroesophageal reflux disease or similar diseases of the stomach, esophagus or digestive tract are providing the most benefit including the long-term effects of treatment (or no treatment) and the progression of the disease over time.

DETAILED DESCRIPTION:
All patients in this registry will have a diagnosis of gastroesophageal reflux disease or a similar disease of the stomach, esophagus or digestive tract. Each patient undergoing anti-reflux surgery will be asked to participate in the registry to gather preoperative, intraoperative and postoperative outcomes. The data collected from the registry will be used to assess the outcome of various treatments, both standard and new: some specific areas of interest include the long-term effects of treatment (or no treatment), the progression of the disease over time, and the overall length of survival of the patient.

ELIGIBILITY:
Inclusion Criteria:

- Any patient undergoing anti-reflux surgery

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of GERD or a similar disease of the stomach, esophagus or digestive tract.
Sampling Method: Non-Probability Sample
Enrollment: 744 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2024-09 (Actual); Study Completion 2024-09 (Actual)

PRIMARY OUTCOMES:
Postoperative patient reported sign and symptoms | Up to 10 years after surgery
  Patient reported signs and symptoms as reported in Reflux scale and GERD questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Leeds, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor Research University Medical Center, Dallas, Texas, United States